CLINICAL TRIAL: NCT00454688
Title: A 12-Week, Randomized, Double-Blind, Dose-Ranging, Placebo-Controlled Study of Asimadoline in Subjects With Irritable Bowel Syndrome
Brief Title: Asimadoline for the Treatment of Subjects With Irritable Bowel Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tioga Pharmaceuticals (Industry)
Collaborators: RTI Health Solutions (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASMP2003
Record Dates: First submitted 2007-03-29; First posted 2007-04-02 (Estimated); Last update posted 2011-10-18 (Estimated); Status verified 2011-10

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome; Asimadoline
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — asimadoline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Asimadoline 0.15 mg (Experimental)
  Interventions: Drug: Asimadoline
- Asimadoline 0.5 mg (Experimental)
  Interventions: Drug: Asimadoline
- Asimadoline 1.0 mg (Experimental)
  Interventions: Drug: Asimadoline

INTERVENTIONS:
Drug: Asimadoline — Asimadoline was provided in coated tablets of three dosages (0.15 mg, 0.5 mg, and 1.0 mg). All asimadoline tablets used in this trial were synthesized from the same batch of drug substance (Batch EF418492). Asimadoline was administered orally, BID for 12 weeks
  Other Names: EMD 61753; EMR 63320
  Arms: Asimadoline 0.15 mg; Asimadoline 0.5 mg; Asimadoline 1.0 mg
Drug: Placebo — Placebo was provided in coated tablets identical in appearance to asimadoline tablets.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of different doses of asimadoline in the treatment of patients with irritable bowel syndrome.

DETAILED DESCRIPTION:
A randomized, dose-ranging, double-blind, placebo-controlled study designed to evaluate the efficacy and tolerability of three dose levels of asimadoline in subjects with IBS.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18-79
* Must sign an ICF
* Females of childbearing potential must have a negative pregnancy test at screening and must adhere to contraception throughout the trial
* Must have been diagnosed with IBS as a result of having at least 6 months, not necessarily consecutive, in the preceding 12 months of recurrent symptoms of abdominal discomfort or pain associated with at least 2 of the following: 1)relieved with defecation; 2)onset associated with a change in stool frequency; 3)onset associated with a change in stool form
* Must demonstrate a willingness to comply with daily telephone diary entry

Exclusion Criteria:

* Any subject with evidence of a biochemical or structural abnormality of the digestive tract or other co-morbid illness that might impact the ability to interpret the safety and efficacy data
* Pregnant or breastfeeding females
* Refusal to discontinue prohibited concomitant medications
* Use of an investigational drug or participation in an investigational study within 30 days of screening
* Inability or unwillingness to use the touch-tone telephone data entry system

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 596 (Actual)
Dates: Start 2006-08; Primary Completion 2007-11 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Relief of IBS Pain - total months | 12 weeks
  The primary efficacy endpoint of the study was the total number of months with adequate relief of IBS pain or discomfort.

SECONDARY OUTCOMES:
Relief of IBS Pain - percent of patients | 12 weeks
  Proportion of subjects with adequate relief of IBS pain or discomfort
Relief of IBS Symptoms | 12 weeks
  Adequate relief of IBS symptoms
Lower GI function - change from baseline | 12 weeks
  Change from baseline in assessments of lower gastrointestinal (GI) function (i.e., stool frequency, stool consistency, urgency, bloating, and straining)
Abdominal Pain Score - change from baseline | 12 weeks
  Change from baseline in abdominal pain score
Abdominal Discomfort Score - change from baseline | 12 weeks
  Change from baseline in abdominal discomfort score

CONTACTS AND LOCATIONS:
Overall Officials: Allen Mangel, MD, PhD, Study Chair — Tioga Pharmaceuticals
Locations (112):
- United States (112):
  - Medical Affiliated Research Center, Huntsville, Alabama
  - Lovelace Scientific Resources, Pheonix, Arizona
  - Lovelace Scientific Resources, Phoenix, Arizona
  - Redpoint Research, Phoenix, Arizona
  - Mayo Clinic Scottsdale - Division of Gastroenterology, Scottsdale, Arizona
  - Genova Clinical Research, Tucson, Arizona
  - Arkansas Gastroenterology, North Little Rock, Arkansas
  - Sutter Institute for Medical Research, Elk Grove, California
  - Digestive & Liver Disease Specialists, Garden Grove, California
  - Irvine Center for Clinical Research Inc., Irvine, California
  - Community Clinical Trials, Orange, California
  - Sutter Institute for Medical Research, Sacramento, California
  - Nothern California Research, Sacramento, California
  - Westlake Medical Research, Westlake Village, California
  - Lynn Institute of the Rockies, Colorado Springs, Colorado
  - Longmont Medical Research Network, Longmont, Colorado
  - Western States Clinical Research Inc, Wheat Ridge, Colorado
  - Clinical Research Consultants, LLC, Stratford, Connecticut
  - Phoenix Internal Medicine Associates, LLC, Waterbury, Connecticut
  - Meridian Research, Brooksville, Florida
  - Florida Medical Research Institute, Gainesville, Florida
  - Research Consultants Group, Hialeah, Florida
  - Suncoast Clinical Research, New Port Richey, Florida
  - Universal Clinical Research & Technology, Orlando, Florida
  - Penninsula Research, Inc, Ormond Beach, Florida
  - Radiant Research - St. Petersburg, Pinellas Park, Florida
  - Lovelace Scientific Resources, Sarasota, Florida
  - Meridien Research, St. Petersburg, Florida
  - Meridien Research, Tampa, Florida
  - Michael S. Levine, MD, Marietta, Georgia
  - Mount Vernon Clinical Research, Sandy Springs, Georgia
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Northwest Gastroenterologists S.C., Arlington Heights, Illinois
  - Illinois Center for Clinical Research, Chicago, Illinois
  - University Digestive Health Center, Oak Forest, Illinois
  - BHS Digestive Disease Associates, Riverside, Illinois
  - Rockford Gastroenterology Associates Ltd, Rockford, Illinois
  - Indianapolis Gastroenterology Research Foundation, Indianapolis, Indiana
  - Heartland Medical Research, Inc, Clive, Iowa
  - Professional Research Network of Kansas, Wichita, Kansas
  - Heartland Research Associates, LLC, Wichita, Kansas
  - University of Louisville GI Research, Louisville, Kentucky
  - Commonwealth Biomedical Research, LLC, Madisonville, Kentucky
  - Digestive Health Center of Louisianna, Baton Rouge, Louisiana
  - Digestive Disorders Associate, Annapolis, Maryland
  - Woodholme Gastroenterology Associates, PA, Baltimore, Maryland
  - Digestive Diseases Associates, PA, Baltimore, Maryland
  - Chevy Chase Clinical Research MGG, Chevy Chase, Maryland
  - Clinical Associates Research, Reisterstown, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Northeast Medical Research Associates, North Dartmouth, Massachusetts
  - Ridgeview Research, Chaska, Minnesota
  - Gastrointestinal Associates, PA, Jackson, Mississippi
  - Olive Branch Family Medical Center, Olive Branch, Mississippi
  - St. Louis Center for Clinical Research, St Louis, Missouri
  - Montana Health Research Institute, Billings, Montana
  - Gastroenterology Specialties, PC, Lincoln, Nebraska
  - Dr. Meera Dewan, PC, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - New Mexico Clinical Research & Osteoporosis Center, Albuquerque, New Mexico
  - Long Island Clinical Research Associates, Great Neck, New York
  - Cornell Weill Medical College, New York, New York
  - Asheville Gastroenterology Associates, PA, Asheville, North Carolina
  - Cary Medical Research Associates, Cary, North Carolina
  - UNC Chapel Hill, Chapel Hill, North Carolina
  - Charlotte Gastroenterology and Hepatology, Charlotte, North Carolina
  - Metrolina Medical Research, Charlotte, North Carolina
  - Cumberland Research Associates, Fayetteville, North Carolina
  - LeBauer research Associates, PA, Greensboro, North Carolina
  - Unifour Medical Research Associates, Hickory, North Carolina
  - Triangle Medical Research Associates, Raleigh, North Carolina
  - Crescent Medical Research, Salisbury, North Carolina
  - Hanover Medical Specialists, PA, Wilmington, North Carolina
  - New Hannover Medical Research, Wilmington, North Carolina
  - Piedmont Medical Research Associates, Winston-Salem, North Carolina
  - Akron Gastroenterology Assoc, Inc., Akron, Ohio
  - Digestive Health Network, Cincinnati, Ohio
  - Radiant Research, Cincinnati, Ohio
  - Radiant Research, Columbus, Ohio
  - Wells Institute for Health Awareness, Kettering, Ohio
  - Radiant Research - Akron, Mogadore, Ohio
  - Lion Research, Norman, Oklahoma
  - Oklahoma Foundation for Digestive Research, Oklahoma City, Oklahoma
  - Options Health Research, LLC, Tulsa, Oklahoma
  - Castlerock Clinical Research Consultants, LLC, Tulsa, Oklahoma
  - NW Gastroenterology Clinic, Portland, Oregon
  - West Hills Gastroenterology Associates, PC, Portland, Oregon
  - Allegheny Center for Digestive Health, Pittsburgh, Pennsylvania
  - Guthrie Clinical Research, Sayre, Pennsylvania
  - Safe Harbor Clinical Research, East Providence, Rhode Island
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Palmetto Medical Research, Mt. Pleasant, South Carolina
  - Hillcrest Clinical Research, Simpsonville, South Carolina
  - ClinSearch, Chattanooga, Tennessee
  - Alpha Clinical Research,LLC, Clarksville, Tennessee
  - Memphis Gastroenterology Group, Germantown, Tennessee
  - Gastroenterology Associates, Kingsport, Tennessee
  - Dial Research Associates, Inc, Nashville, Tennessee
  - Covance CRU-Austin, Austin, Texas
  - Sadler Clinic, Conroe, Texas
  - Texas Tech University Health Sciences Center, El Paso, Texas
  - Discovery Alliance, Houston, Texas
  - NationsMed Clinical Research, Houston, Texas
  - Clinical Trials Network, Houston, Texas
  - Texas Tech University Health Sciences Center, Lubbock, Texas
  - Sun Research Institute, San Antonio, Texas
  - Advanced Research Institute, Ogden, Utah
  - J. Lewis Research Inc., Foothills Family Clinic, Salt Lake City, Utah
  - Charlottesville Medical Research, Charlottesville, Virginia
  - New River Valley Research Institute, Christiansburg, Virginia
  - National Clinical Research Inc, Richmond, Virginia
  - Wisconsin Center for Advanced Research, Milwaukee, Wisconsin